CLINICAL TRIAL: NCT00295906
Title: Efficacy of Web-Based Instruction on Skin Cancer Triage
Brief Title: Computer-Based Continuing Education for Doctors in Examination and Counseling of Patients on Skin Cancer or Weight Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized
Other Study IDs: CDR0000454721; RIH-1050258954A1; RIH-0348-03
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2008-11

CONDITIONS: Melanoma (Skin); Non-melanomatous Skin Cancer
Keywords: melanoma; skin cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Early Intervention, Educational

INTERVENTIONS:
Other: educational intervention
Other: internet-based intervention

SUMMARY:
RATIONALE: Computer-based continuing education courses may be effective in improving the skills of primary care doctors to identify skin cancer risk factors, perform skin cancer exams, and counsel patients. They may also improve the skills of primary care doctors to assess and counsel patients on their weight, diet, and physical activity.

PURPOSE: This randomized clinical trial is studying how well computer-based continuing education courses work in improving doctors' ability to perform skin cancer or weight control exams and counseling during routine office visits.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of a continuing education course designed to improve primary care physician performance in examination and counseling of patients about skin cancer vs a continuing education course designed to improve physician assessment of weight management.
* Evaluate physician performance of skin examination during routine patient visits at 12 months after completion of the skin cancer continuing education course.
* Evaluate physician counseling around skin cancer issues.

Secondary

* Evaluate the efficacy of the skin cancer continuing education course in improving physician skin cancer triage skills and in changing physician attitudes and knowledge regarding skin cancer issues.
* Assess improvements in physician assessment of weight, diet, and physical activity.

OUTLINE: This is a randomized, multicenter study. Physicians are stratified according to participating center. Physicians are randomized to 1 of 2 intervention arms.

* Arm I (skin cancer continuing education course): Physicians complete a 1-hour continuing education course on skin cancer. The course is available to the physician as a reference for up to 12 months. Physicians complete an online test at baseline, immediately after the course is completed, and at 1 month and 12 months after course completion to assess their knowledge, attitudes, skill, and practices towards skin examination and skin cancer counseling.

Patients are interviewed by telephone within 1 week after a routine office visit with their physician to assess the physician's skin assessment and skin cancer counseling practices. The interviews are conducted prior to and at 1 month and 12 months after the physician completes the continuing education course.

* Arm II (weight control continuing education course): Physicians complete a 1-hour continuing education course on weight, dietary, and physical activity assessment and counseling. The course is available to the physician as a reference for up to 12 months. Physicians complete an online test at baseline, immediately after the course is completed, and at 1 month and 12 months after course completion to assess their knowledge, attitudes, skill, and practices towards weight, dietary, and physical activity assessment and counseling.

Patients are interviewed by telephone within 1 week after a routine office visit with their physician to assess the physician's weight, dietary, and physical activity assessment and counseling practices. The interviews are conducted prior to and at 1 month and 12 months after the physician completes the continuing education course.

PROJECTED ACCRUAL: A total of 50 physicians and 4,500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Primary care physician, meeting all of the following criteria:

  * General internist or family physician
  * Must devote at least 75% of their time to primary care practice
  * At least 1 year in practice
  * Must be in a community-based practice with no more than 1 participating physician per practice
  * Must not be planning to retire within the next 2 years
  * Has a patient population that is predominantly at substantial risk of melanoma and other skin cancers (i.e., adults whose non-sun-exposed skin color is white or tan, but not brown)
* Patient

  * Adult who is scheduled for a routine office visit with a study physician

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4550 (Estimated)
Dates: Start 2004-06; Primary Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Patient exit interviews at 12 months

SECONDARY OUTCOMES:
Patient exit interviews at 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin A. Weinstock, MD, PhD, Study Chair — Rhode Island Hospital
Locations (5):
- United States (5):
  - Scripps-Ranch Family Medicine Clinic at University of California, San Diego, California
  - University of Kansas School of Medicine - Wichita, Wichita, Kansas
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island